CLINICAL TRIAL: NCT06628557
Title: "The Effect of Mandala Art Therapy on Anxiety and Pain in Patients Undergoing Total Hip Replacement: A Randomized Controlled Study"
Brief Title: The Effect of Mandala Art Therapy on Anxiety and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seval Ulubay (Other)
Responsible Party: Sponsor-Investigator, Seval Ulubay, PhD, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mandala Art
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Total Hip Replacement
Keywords: The Effect of Mandala Art Therapy; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study aims to evaluate the effects of mandala art therapy on anxiety and pain in patients undergoing total hip replacement. The data obtained from the research is expected to provide evidence regarding the impact of mandala art therapy, a non-pharmacological approach, on anxiety and pain levels in post-operative patients who have undergone total hip replacement.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of Mandala Art Therapy on Anxiety in Patients Undergoing Total Hip Replacement (Experimental): Between May 22, 2024, and December 30, 2024, patients undergoing total hip replacement surgery at Samsun Gazi State Hospital's Orthopedic Surgery Clinic will be informed about the study. Between May 22, 2024, and December 30, 2024, patients undergoing total hip replacement surgery at Samsun Gazi State Hospital's Orthopedic Surgery Clinic will be informed about the study. Those who agree to participate will complete an Informed Consent Form, Patient Introduction Form, Pain Assessment Scale, and State-Trait Anxiety Inventory (STAI-I). One group will engage in mandala coloring activities using a coloring book on the second day post-surgery, while the other group will not receive this intervention. The same questionnaires will be administered again after the intervention.
  Data Analysis Data evaluation will utilize frequency, percentage, mean, standard deviation, Student's t-test, analysis of variance, and Pearson correlation analysis.
  Interventions: Other: The Effect of Mandala Art Therapy on Anxiety and Pain in Patients
- The Effect of Mandala Art Therapy on Pain in Patients Undergoing Total Hip Replacement (Experimental): Between May 22, 2024, and December 30, 2024, patients undergoing total hip replacement surgery at Samsun Gazi State Hospital's Orthopedic Surgery Clinic will be informed about the study. Between May 22, 2024, and December 30, 2024, patients undergoing total hip replacement surgery at Samsun Gazi State Hospital's Orthopedic Surgery Clinic will be informed about the study. Those who agree to participate will complete an Informed Consent Form, Patient Introduction Form, Pain Assessment Scale, and State-Trait Anxiety Inventory (STAI-I). One group will engage in mandala coloring activities using a coloring book on the second day post-surgery, while the other group will not receive this intervention. The same questionnaires will be administered again after the intervention.
  Data Analysis Data evaluation will utilize frequency, percentage, mean, standard deviation, Student's t-test, analysis of variance, and Pearson correlation analysis.
  Interventions: Other: The Effect of Mandala Art Therapy on Anxiety and Pain in Patients

INTERVENTIONS:
Other: The Effect of Mandala Art Therapy on Anxiety and Pain in Patients — The Effect of Mandala Art Therapy on Anxiety and Pain in Patients
  Other Names: The Effect of Mandala Art Therapy

SUMMARY:
This study aims to evaluate the effects of mandala art therapy on anxiety and pain in patients undergoing total hip replacement. The data obtained from the research is expected to provide evidence regarding the impact of mandala art therapy, a non-pharmacological approach, on anxiety and pain levels in post-operative patients who have undergone total hip replacement.

DETAILED DESCRIPTION:
Hip arthroplasty is recognized as an effective method for adults suffering from significant pain and limited mobility due to hip joint damage. The rapid advancements in total hip arthroplasty technology, alongside the increasing average life expectancy, highlight the importance of this procedure for patients who have undergone it. However, any surgical intervention can be traumatic for patients. Experiencing surgical trauma often leads to pain, and approximately 60-80% of individuals exhibit anxiety prior to such procedures. Factors contributing to anxiety and pain are frequently linked to a person's emotional, psychological, behavioral, and socio-cultural background. Previous studies have emphasized that anxiety and pain behaviors, which can adversely affect individuals during surgical processes, are related to the perception of pain. Effective and planned nursing care can significantly reduce pre-operative anxiety, resulting in lower levels of pain and anxiety post-surgery. In patients undergoing total hip arthroplasty, it is essential to manage post-operative acute pain effectively. Successful pain management allows patients to mobilize more quickly and reduces hospital stay durations. Severe post-operative pain can discourage patients from engaging in necessary exercises. To control this acute pain, it is often recommended to administer analgesics every 4-6 hours, based on medical advice. Regular pain assessment, establishing therapeutic communication with patients, and employing patient-controlled analgesia, along with oral analgesics, are among the most effective pain management strategies. Additionally, non-pharmacological methods are suggested as alternatives to pharmacological approaches. Mandala art therapy represents an inward journey for individuals, helping them feel empowered and extraordinary. The mandala, depicting the blossoming of a flower at its center, symbolizes the spiritual self. While representing unity, the mandala forms a pattern that transitions from the micro to the macro, symbolizing the moment of existence and life. Jung utilized mandala art as a therapeutic method and since then, it has been applied across various fields as mandala therapy. The mandala activity has been associated with positive psychological effects, such as enhancing individual awareness, boosting self-esteem, and reducing feelings of guilt . Literature suggests that engaging with mandalas fosters conscious awareness and positively contributes to individuals. This engagement helps focus attention and distances individuals from negative thoughts, thereby alleviating anxiety. While no significant differences have been observed between mandala coloring and drawing in terms of anxiety reduction, mandala coloring may be preferred in the future for its cost-effectiveness and ease of implementation for adults . One study found that engaging in mandala activities for at least 30 minutes daily significantly reduced anxiety levels in patients, offering an adjunctive treatment option. Another study emphasized that performing mandala activities with focus could positively impact psychological and emotional well-being, thereby reducing anxiety. A systematic meta-analysis indicated that mandala activities significantly and positively affect state anxiety. Reducing pain and anxiety in patients who have undergone total hip replacement will enhance patient comfort and satisfaction. Therefore, this study aims to evaluate the effects of mandala art therapy on anxiety and pain in patients undergoing total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total hip replacement in the orthopedic surgery clinic.
* Patients aged 18 and over.

Exclusion Criteria:

* Patients under the age of 18.
* Patients undergoing total hip replacement surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Surgical Fear Scale | 8 weeks
  A low score on the surgical fear scale indicates a low level of surgical anxiety.
Visual Analog Scale (VAS) | 8 weeks
  It is displayed on a straight line between 0 and 10. As the numerical value increases, so does the stress level.

CONTACTS AND LOCATIONS:
Overall Officials: Seval ULUBAY, PHD, Principal Investigator — Samsun Gazi State Hospital
Locations (1):
- Seval Ulubay, Samsun, Atakum/Samsun, Turkey (Türkiye)